CLINICAL TRIAL: NCT06391177
Title: A Phase 1, Open-label Study to Evaluate Vonoprazan Concentrations in Breast Milk of Healthy Lactating Women Receiving Vonoprazan 20 mg Once Daily or Vonoprazan 20 mg Twice Daily
Brief Title: A Study to Evaluate Vonoprazan Concentrations in Breast Milk of Healthy Lactating Women Receiving Vonoprazan 20 mg Once Daily or Vonoprazan 20 mg Twice Daily
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Phathom Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: VONO-401
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-02

CONDITIONS: Erosive Esophagitis; Heartburn; Symptomatic Nonerosive Gasroesophageal Reflux Disease; Helicobacter Pylori Infection
Keywords: Healthy participants; Helicobacter pylori infection; Erosive Esophagitis; Symptomatic nonerosive gasroesophageal reflux disease; Heartburn; Breast milk; Lactating women
MeSH Terms: conditions — Heartburn | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vonoprazan 20 mg Once Daily (Experimental): Participants will be administered once-daily doses of vonoprazan 20 mg for 4 consecutive days (Days 1 through 4).
  Interventions: Drug: Vonoprazan
- Vonoprazan 20 mg Twice Daily (Experimental): Participants will be administered twice-daily doses of vonoprazan 20 mg for 4 consecutive days (Days 1 through 4).
  Interventions: Drug: Vonoprazan

INTERVENTIONS:
Drug: Vonoprazan — Oral tablet.

SUMMARY:
The primary objective is to determine the pharmacokinetics (PK) of vonoprazan in breast milk of healthy lactating women who have received vonoprazan administered once daily or vonoprazan 20 mg administered twice daily for 4 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is a healthy lactating woman at least 18 years of age at the time of signing the informed consent form (ICF).
2. The participant has delivered a normal term infant (at least 37 weeks gestation) and has been breastfeeding or actively pumping breast milk for at least 4 weeks postpartum prior to the first dose.
3. The participant is willing to not breastfeed or otherwise use her breast milk during administration of vonoprazan and until at least 5 days after the last dose of the study drug.
4. The participant has confirmed that her breastfed infant is able to feed from a bottle.
5. The participant agrees to collect all breast milk from pre-dose to 24 hours after the morning dose administration on Day 4, using an electric pump.
6. The participant is considered by the investigator to be in good general health as determined by medical history, clinical laboratory test results, vital sign measurements, 12-lead ECG results, and physical examination findings at Screening.
7. Participants of childbearing potential must use an acceptable method of birth control (ie, diaphragm with spermicide, intrauterine device, condom with foam or vaginal spermicide, oral contraceptives, or abstinence) or be surgically sterile (ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy). All participants must have a negative pregnancy test at Screening and before the first dose of study drug (Baseline).
8. The participant agrees to comply with all protocol requirements.
9. The participant is able to provide written informed consent.

Exclusion Criteria:

1. The participant has a positive pregnancy test at Screening or Baseline, is planning to become pregnant before, during, or within 4 weeks after participating in this study, or intends to donate ova during this time period, or is of childbearing potential and not using an effective contraceptive method.
2. The participant has a history of breast implants, breast augmentation, or breast reduction surgery that significantly impacts breastfeeding or collection of milk from one or both breasts.
3. The participant has signs or symptoms of mastitis or other condition that would prevent the collection of milk from one or both breasts.
4. The participant has undergone prior esophageal and/or gastrointestinal surgeries that may affect study drug absorption.
5. The participant has undergone surgery (other than cesarean section) within 30 days before the first dose of study drug.
6. The participant has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus types 1 or 2 antibodies at Screening.
7. The participant has any other clinically significant findings on physical examination, clinical laboratory abnormalities, or ECG results that preclude participation in the study, as deemed by the investigator.
8. The participant has used any prescription (excluding hormonal birth control) and/or over-the-counter medications (including cytochrome P450 3A4 inducers), including herbal or nutritional supplements, within 14 days before the first dose of study drug, and/or is expected to require any such medication during the course of the study until end of the Treatment Period. Use of multivitamins and acetaminophen (up to 2 g per day) is permissible.
9. The participant has consumed grapefruit and/or grapefruit juice, Seville orange, or Seville orange-containing products (eg, marmalade) within 7 days before the first dose of study drug and/or is expected to be unable to abstain through the study.
10. The participant is a smoker or has used nicotine or nicotine-containing products (eg, snuff, nicotine patch, nicotine chewing gum, mock cigarettes, or inhalers) within 6 months before the first dose of study drug.
11. The participant has a history of alcohol abuse or drug dependency within 12 months before the first dose of study drug.
12. The participant has a positive test result for drugs of abuse, alcohol, or cotinine (indicating active current smoking) at Screening, Baseline, or Day 4 (Check-in).
13. The participant is involved in strenuous activity or contact sports within 24 hours before the first dose of study drug and during the study.
14. The participant has a history of relevant drug and/or food allergies (ie, any significant food allergy that could preclude a standard diet in the clinical research unit).
15. The participant has received study drug in another investigational study (including vonoprazan) within 30 days prior to start of the Screening Period.
16. The participant has a history of hypersensitivity or allergies to vonoprazan or any of its formulation excipients (D-mannitol, microcrystalline cellulose, hydroxypropyl cellulose, fumaric acid, ascorbic acid, croscarmellose sodium, magnesium stearate, hypromellose, polyethylene glycol 8000, titanium dioxide, or ferric oxide red).
17. In the opinion of the investigator, the participant is not suitable for entry into the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Development, LP, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 15 participants were enrolled in the United States between May 2024 and September 2024.
Pre-assignment Details: Participants were administered vonoprazan once daily (QD) or twice daily (BID).
Groups:
- Vonoprazan 20 mg QD: Participants were administered vonoprazan 20 mg QD for 4 consecutive days (Days 1 through 4).
- Vonoprazan 20 mg BID: Participants were administered vonoprazan 20 mg BID for 4 consecutive days (Days 1 through 4).
Period: Overall Study
Arm/Group | Vonoprazan 20 mg QD | Vonoprazan 20 mg BID
Started | 5 | 10
Completed | 5 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population: included all participants who received at least 1 dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vonoprazan 20 mg QD | Vonoprazan 20 mg BID | Total
Number analyzed (Participants) | 5 | 10 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.4 (4.45) | 29.7 (3.71) | 31.3 (4.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 4 | 10 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 8 | 12
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under Drug Concentration-time Curve From Time 0 to 24 Hours (AUC0-24) Following the Morning Dose of Vonoprazan in Breast Milk
Description: AUC from time 0 to 24 hours post-dose, calculated as: the sum of the product of the concentration of the interval and the width of the interval.
Time Frame: Pre-dose on Day 4, and at regularly scheduled intervals through 24 hours after the morning dosing (0-4 hours, 4-8 hours, 8-12 hours, 12-18 hours, and 18-24 hours).
Population: PK population: included all participants who received sufficient doses of vonoprazan and had sufficient concentration data in milk to support accurate estimation of at least 1 PK parameter in milk.
Measure: Mean (Standard Deviation); unit: ng•h/mL
Arm/Group | Vonoprazan 20 mg QD | Vonoprazan 20 mg BID
Number analyzed (Participants) | 5 | 10
ng•h/mL | 179 (61.3) | 317 (107)

2. Primary Outcome: Maximum Drug Concentration (Cmax) of Vonoprazan in Breast Milk
Description: Maximum observed concentration after dosing.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vonoprazan 20 mg QD | Vonoprazan 20 mg BID
Number analyzed (Participants) | 5 | 10
ng/mL | 20.9 (6.02) | 24.7 (9.77)

3. Primary Outcome: Minimum Drug Concentration (Cmin) of Vonoprazan in Breast Milk
Description: Minimum observed concentration after dosing.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vonoprazan 20 mg QD | Vonoprazan 20 mg BID
Number analyzed (Participants) | 5 | 10
ng/mL | 1.82 (0.833) | 6.78 (2.19)

4. Primary Outcome: Average Drug Concentration (Cavg) of Vonoprazan in Breast Milk
Description: Average concentration, calculated as: AUC0-24/tau (tau=the difference between the end time of the last interval and dosing time).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vonoprazan 20 mg QD | Vonoprazan 20 mg BID
Number analyzed (Participants) | 5 | 10
ng/mL | 7.55 (2.58) | 13.3 (4.51)

5. Primary Outcome: Time to Cmax (Tmax) of Vonoprazan in Breast Milk
Description: Time to maximum observed concentration (actual midpoint of the interval in which Cmax was observed).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Vonoprazan 20 mg QD | Vonoprazan 20 mg BID
Number analyzed (Participants) | 5 | 10
hours | 1.88 [1.83 to 1.93] | 1.91 [1.88 to 14.8]

6. Secondary Outcome: Total Amount of Vonoprazan Excreted in Breast Milk
Description: Total amount of drug excreted in breast milk over 24 hours; calculated as the sum of drug concentration × expressed milk volume in each collection interval over 24-hour period.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Vonoprazan 20 mg QD | Vonoprazan 20 mg BID
Number analyzed (Participants) | 5 | 10
mg | 0.00241 (0.00118) | 0.00904 (0.00530)

7. Secondary Outcome: Percentage of Vonoprazan Excreted in Breast Milk Relative to the Total Dose Received
Description: Total amount of drug excreted over 24 hours relative to total dose administered; calculated as the sum of (total amount of drug excreted in each collection interval / total dose received over 24-hour period) * 100.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of vonoprazan
Arm/Group | Vonoprazan 20 mg QD | Vonoprazan 20 mg BID
Number analyzed (Participants) | 5 | 10
percentage of vonoprazan | 0.0120 (0.00592) | 0.0226 (0.0132)

8. Secondary Outcome: Estimated Infant Daily Dose of Vonoprazan
Description: Estimated weight adjusted daily dose consumed by the infant through breast milk; calculated as total amount of drug excreted over 24-hour period / weight of infant.
  Calculation used the nominal infant weight of 6.0 kg which is the approximate 50th percentile for a 3-month old infant.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/kg/day
Arm/Group | Vonoprazan 20 mg QD | Vonoprazan 20 mg BID
Number analyzed (Participants) | 5 | 10
mg/kg/day | 0.000401 (0.000197) | 0.00151 (0.000883)

9. Secondary Outcome: Estimated Relative Infant Dose to the Total Maternal Dose Received of Vonoprazan
Description: Percentage of daily infant dose relative to the daily maternal dose; calculated as (daily infant dose / daily maternal dose) * 100.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of total maternal dose
Arm/Group | Vonoprazan 20 mg QD | Vonoprazan 20 mg BID
Number analyzed (Participants) | 5 | 10
percentage of total maternal dose | 0.128 (0.0556) | 0.269 (0.186)

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 11
Description: A treatment emergent adverse event (TEAE) was defined as any event that occurred after the first dose of the study drug or any event at Baseline that worsened in either intensity or frequency after the first dose of the study drug until 30 days after the last dose of the study drug.
  Safety population: included all participants who received at least 1 dose of study drug.
Arm/Group | Vonoprazan 20 mg QD | Vonoprazan 20 mg BID
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/10
Other Adverse Events (participants affected / at risk) | 1/5 | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vonoprazan 20 mg QD (N=5) | Vonoprazan 20 mg BID (N=10)
Nausea (Gastrointestinal disorders) | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigators (PIs) are not permitted to publish the data. Data may be considered for reporting at a scientific meeting or for publication in a scientific journal. In these cases, the sponsor will be responsible for these activities and will work with the PIs to determine how the manuscript is written and edited, the number and order of authors, the publication to which it will be submitted, and any other related issues. The sponsor has final approval authority over all such issues.

DOCUMENTS (2):
  • Study Protocol (2024-07-18): https://cdn.clinicaltrials.gov/large-docs/77/NCT06391177/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-30): https://cdn.clinicaltrials.gov/large-docs/77/NCT06391177/SAP_001.pdf